CLINICAL TRIAL: NCT02123836
Title: Pilot Study of Expanded, Activated Haploidentical Natural Killer Cell Infusions for Non-B Lineage Acute Leukaemia and Myelodysplastic Syndrome
Brief Title: Natural Killer Cells in Acute Leukaemia and Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKEXPSIN-2013/01
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Acute Leukaemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NK cells (Experimental): Peripheral blood cell will be collected by apheresis from donors. Peripheral blood mononucleated cells will be cultured with irradiated K562-mb15-41BBL cells and low dose (10 IU/mL) IL-2 for 10 days. After T-cell depletion, expanded activated NK cells will be infused. Before infusion, patients will receive immunosuppressive therapy to promote temporary engraftment of NK cells. After infusion, they will receive IL-2 to support NK cell viability and expansion in vivo. The effects of NK cell infusion will be determine by comparing MRD levels before and after treatment.
  Interventions: Biological: NK cells

INTERVENTIONS:
Biological: NK cells — 7 days of preparatory treatment are given before the NK cell infusion. Chemotherapy will be given over 6 days. This chemotherapy will promote donor NK cells engraftment. After which, a drug called Interleukin-2 (IL-2) will be given as an injection just under the skin three times per week for at least 2 weeks (total of 6 doses). This treatment is used to help keep the donor NK cells alive.
  Blood cells will be collected from an eligible and suitable family donor 10 days before infusion. The collection sample will be processed to remove red blood cells and as many T-cells as possible. T-cells from the donor might cause these donor cells to attack the body, usually the skin, liver, and intestines.
  NK cells will be activated in the National University Hospital lab and ready for infusion on Day 0.
  The NK cells will then be infused into the vein, through a peripheral catheter.

SUMMARY:
A novel method has been developed to expand natural (NK) cells and enhance their cytotoxicity against cancer cells while maintaining low killing capacity against non-transformed cells. In this method, donor NK cells are expanded by co-culture with the irradiated K562 cell line modified to express membrane bound IL-15 and 41BB ligand (K562-mb15-41BBL). Expression of these proteins in conjunction with unknown stimuli provided by K562 cells promotes selective growth of NK cells. Then, the expanded NK cell population is depleted of T cells to prevent graft versus host disease (GVHD). Expanded and activated NK cells showed powerful anti-leukemic activity against acute myeloid leukemia (AML) cells in vitro and in animal models of leukemia.Unpublished laboratory results also demonstrated that T-cell acute lymphoblastic leukaemia (T-ALL) is extremely sensitive to the cytotoxicity exerted by the expanded and activated NK cells.

The present study represents the translation of the laboratory findings into clinical application. The study proposes to determine the feasibility, safety and efficacy of infusing expanded NK cells into patients who have AML or T-lineage ALL which is resistant to standard therapy as demonstrated by persistent minimal residual disease (MRD). Patients with myelodysplastic syndrome (MDS), who are at high risk to develop AML will also be eligible for the study. In this patient cohort, the study will also investigate the in vivo lifespan and phenotype of the expanded NK cells.

The main hypothesis to be tested in this study is that infusion of expanded activated NK cells can produce measurable clinical responses in patients with AML or T-ALL.

DETAILED DESCRIPTION:
The study will enroll 20 eligible subjects who will receive NK cell infusion to test whether infusion of expanded activated NK cells can produce measurable clinical responses in patients with AML/MDS or T-ALL.The study aims to infuse a target dose of 10 x 107 CD56+ cells/kg, however, as the actual cell dose obtained will vary depending on the donor harvest, the accepted range for cell infusion will be 0.5-20 x 107 CD56+ cells/kg. On day -10, eligible donors (adult family member of recipient) will undergo apheresis once. A second apheresis procedure may be needed to obtain the required cell count from the donor. NK cells will be expanded in co-culture with irradiated (100 Gy) K562-mb15-41BBL cells in closed culture containers for 10 days. Prior to NK cell infusion on Day 0, recipients will undergo screening evaluations and will receive cyclophosphamide, Fludarabine, IL-2, and supportive medications (e.g. mesna). Cytokine regimen of IL-2 will be initiated on the evening of day -1 (dose 1 of 6). IL-2 will be continued at a dose of 1 million units/m2 subcutaneously 3 times per week for 2 weeks (6 doses total). Post-infusion follow-up procedures for up to 1 year from the day of NK cell infusion include physical examination, Complete Blood Count, and metabolic/chemistry studies. The effects of NK cell infusion will also be determined by comparing MRD levels before and after treatment. MRD blood and bone marrow levels will be collected at baseline and at specified time points (until 1 year from the day of NK cell infusion). NK cell donors will be recruited from the family members of the patient recipient. Potential donors aged 21 years old will be consented and will undergo the required screening tests and human leukocyte antigen (HLA) typing. Since 20 eligible subjects will be enrolled as NK cell recipients, 20 donors will also be recruited for this study. Ineligible NK cell donors will have to be replaced.

ELIGIBILITY:
Inclusion Criteria: (NK cell Recipient)

* From 6 to 80 years old at time of consent.
* Patients with the following haematological diseases:

  * Acute myeloid leukaemia (de novo or secondary)
  * Myelodysplastic syndromes (RAEB I/II)
  * T-cell acute lymphoblastic leukaemia (T-ALL)
* Patients must have been treated with prior standard intensive chemotherapy upfront, which will be defined according to institutional practice for each respective disease, and may include allogeneic haematopoietic stem cell transplantation.
* Patients must have persistent detectable residual leukaemia following initial treatment with intensive chemotherapy. Residual leukaemia is defined as the presence of >=0.01%-20% blasts in the bone marrow by flow cytometry.

  * High risk AML patients with either High risk cytogenetics or FLT3-ITD mutation or Acute megakaryoblastic leukaemia in non-Down's Therapy related leukaemia or Myelodysplastic syndrome

will qualify for NKEXPSIN either after Induction I chemotherapy or Induction II chemotherapy regardless of residual disease.

* At least two weeks since receipt of any biological therapy, chemotherapy, and/or radiation therapy.
* Shortening fraction greater than or equal to 25%.
* Glomerular filtration rate greater than or equal to 60ml/min.
* Pulse oximetry greater than or equal to 92% on room air.
* Direct bilirubin less than or equal to 3x Upper Limit of Normal (ULN).
* Karnofsky performance score of greater than or equal to 50.
* Has a suitable adult family member donor available for NK cell donation.
* Ability to provide informed consent. Otherwise, a legally authorized representative (LAR) must be present throughout the consent process and is allowed to give consent on the patient's behalf.

Inclusion Criteria: (NK cell Donor)

* At least 21 years old at time of consent.
* A family member with a greater than or equal to 3 of 6 HLA match to recipient
* Ability to provide informed consent. Otherwise, a legally authorized representative must be present throughout the consent process and is allowed to give consent on the patient's behalf.

Exclusion Criteria: (NK cell Recipient)

* Currently has pleural or pericardial effusion.
* Receiving more than the equivalent of prednisone 10 mg daily.
* Lactating or pregnant. Negative serum or urine pregnancy test result must be within 7 days prior to enrolment.

Exclusion Criteria: (NK cell Donor)

* HIV positive. Negative results must be within 60 days prior to enrolment.
* Lactating or pregnant. Negative serum or urine pregnancy test result must be within 7 days prior to enrolment.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD) levels | 1 year
  MRD blood levels will be tested at baseline, weekly during the first 2 months and monthly thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Frances Yeap, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Fujisaki H, Kakuda H, Shimasaki N, Imai C, Ma J, Lockey T, Eldridge P, Leung WH, Campana D. Expansion of highly cytotoxic human natural killer cells for cancer cell therapy. Cancer Res. 2009 May 1;69(9):4010-7. doi: 10.1158/0008-5472.CAN-08-3712. Epub 2009 Apr 21. PMID 19383914
- [Background] Imai C, Iwamoto S, Campana D. Genetic modification of primary natural killer cells overcomes inhibitory signals and induces specific killing of leukemic cells. Blood. 2005 Jul 1;106(1):376-83. doi: 10.1182/blood-2004-12-4797. Epub 2005 Mar 8. PMID 15755898
- [Background] Fujisaki H, Kakuda H, Imai C, Mullighan CG, Campana D. Replicative potential of human natural killer cells. Br J Haematol. 2009 Jun;145(5):606-13. doi: 10.1111/j.1365-2141.2009.07667.x. Epub 2009 Mar 26. PMID 19344420
- See also: National University Cancer Institute, Singapore — http://www.ncis.com.sg/